

# İNÖNÜ ÜNİVERSİTESİ SAĞLIK BİLİMLERİ BİLİMSEL ARAŞTIRMA VE YAYIN ETİĞİ BİLGİLENDİRİCİ GÖNÜLLÜ ONAM FORMU



# THE EFFECT OF THERAPEUTIC TOUCH AND MUSIC REST ON SLEEPING APPLIED TO CHILDREN WITH LIVER TRANSPLANTATION

ID: TDK-2020-2358

NCT ID not yet assigned

Initial Release: 09/09/2021

You Assoc. Dr. We invite you to the research titled "The Effects of Therapeutic Touch and Music Concert for Children with Liver Transplantation" conducted by Maksude YILDIRIM under the consultancy of Emriye Hilal YAYAN. Before deciding whether or not to participate in this research, you need to know why and how the research will be conducted. Therefore, it is very important to read and understand this form. If there is something that you do not understand and is not clear to you, or if you want more information, ask us.

Participation in this study is completely voluntary. You have the right not to participate in the study or to withdraw from the study at any time after participating. Participants/Volunteers were informed by making explanations. Required Permission/Consent was obtained for the study. Your participation in the study, answering the questions means that you give your consent / consent to participate in the research. Do not be under pressure or suggestion from anyone while answering the questions on the forms given to you. The information obtained from these forms will be used for research purposes only. Even if the research is published, your name and identity information will remain strictly confidential and will not be given to a third party.

- 1. TITLE OF THE SURVEY: "THE EFFECT OF THERAPEUTIC TOUCH AND MUSIC REST ON SLEEPING APPLIED TO CHILDREN WITH LIVER TRANSPLANTATION"
- **2. NUMBER OF PARTICIPANTS:** The total number of participants envisaged to take part in this study is 50.
- **3. DURATION OF PARTICIPATION IN THE RESEARCH:** The estimated time for you to take part in this research is 5 days.

## 4. OBJECTIVE OF THE RESEARCH:

This research was planned to examine the "The Effects of Therapeutic Touch and Music Rest on Sleeping Applied to Children with Liver Transplantation".



# İNÖNÜ ÜNİVERSİTESİ SAĞLIK BİLİMLERİ BİLİMSEL ARAŞTIRMA VE YAYIN ETİĞİ BİLGİLENDİRİCİ GÖNÜLLÜ ONAM FORMU



## 5. CONDITIONS FOR PARTICIPATION IN THE RESEARCH

The conditions you must meet to be included in this research are as follows;

- \*At least one month and a maximum of two years after the transplant
- \* 0-18 years old
- \* Conscious
- \*spontaneous breathing
- \*No hearing problems
- \*Pain free
- \*Children who do not use sleeping pills will be included in the study.

## 6. METHOD OF THE RESEARCH

# The procedures to be performed in this research are as follows;

The data of the research will be collected by face-to-face interview technique with the "Introductory Information Form", "Actigraphy" created by the researcher between February 2021 and October 2021.

# 7. POTENTIAL RISKS ARISING FROM INVESTIGATION

Necessary measures will be taken by us against a possible problem.

There are no possible risks.

#### 8. LIABILITY / LIABILITY IN CASE OF ANY DAMAGE RESULTING FROM THE RESEARCH

If you suffer any damage as a result of the research, the necessary expenses will be covered by the researchers.

## 9. PERSON TO CALL FOR PROBLEMS THAT MAY OCCUR DURING THE RESEARCH

During the application, you can reach the relevant physician, whose address and phone are given below, at any time to inform the Responsible Investigator in advance if you have to take non-study medication forcibly, to get additional information about the trial, or for any problems, undesirable effects or other discomforts related to the trial.

Address and Telephones of your Researcher, who can be reached 24 hours a day, whenever you want:

İnönü University Faculty of Nursing, Department of Child Health and Diseases Nursing / Malatya **Work:** 0 422 341 02 20 **Mobile:** 0530-324-39-89



# İNÖNÜ ÜNİVERSİTESİ SAĞLIK BİLİMLERİ BİLİMSEL ARAŞTIRMA VE YAYIN ETİĞİ BİLGİLENDİRİCİ GÖNÜLLÜ ONAM FORMU



## CONSENT TO PARTICIPATE IN THE RESEARCH

I have read the above information that should be given to the participant/volunteer before the research and I fully understand the scope and purpose of the study I am asked to participate in, and my responsibilities as a volunteer. Written and verbal explanation about the study was made by the researcher whose name is mentioned below. I had the opportunity to ask questions and discuss and got satisfactory answers. To me; The possible risks and benefits of the study were also explained orally. I understood that I could leave this work whenever I wanted and without having to give any reason, and that I would not face any negative consequences if I quit.

In these circumstances, I agree to participate in the research in question voluntarily, without any pressure or coercion.

| VOLUNTARILY | SIGNATURE/DATE |
|------------------|----------------|
| NAME AND SURNAME | |
| ADDRESS | |
| TELEPHONE | |
| DATE | |

| PARENT/GUARDIAN | SIGNATURE/DATE |
|------------------|----------------|
| NAME AND SURNAME | |
| ADDRESS | |
| TELEPHONE | |
| DATE | |

| ARAŞTIRMACI | | SIGNATURE/DATE |
|---|---|---|
| NAME-SURNAME and POSITION | Maksude YILDIRIM ( Research Assistant ) | |
| ADDRESS | İnönü University Faculty of Nursing, Child Health and Diseases Nursing/Malatya | |
| TELEPHONE | 0530-324-39-89 | |
| DATE | | |